CLINICAL TRIAL: NCT07132333
Title: The Molecular Inflammation Board at the Centers for Personalized Medicine at the University Hospitals of Freiburg, Heidelberg, Tübingen and Ulm - A Multicenter Prospective Observational Study
Brief Title: Molecular Inflammation Board at the Center for Personalized Medicine
Acronym: MEB@ZPM
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Freiburg (Other); University Hospital Heidelberg (Other); University Hospital Ulm (Other)
Responsible Party: Sponsor
Other Study IDs: 482/2022BO1
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis (PsO); Psoriasis Arthritis; Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis); Spondylarthropathies
Keywords: chronic inflammatory diseases; personalized medicine
MeSH Terms: conditions — Psoriasis; Inflammatory Bowel Diseases; Colitis, Ulcerative; Spondylarthropathies | interventions — Biological Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Biologic Agent — Intervention with biologic agents

SUMMARY:
Molecular Inflammation Board at the Center for Personalized Medicine

DETAILED DESCRIPTION:
Molecular Inflammation Board at the Center for Personalized Medicine

The study objectives are:

To ensure a prospective documentation of all patients who are referred to the Molecular Inflammation Board in routine clinical care To prospectively ensure the documentation of MEB patients with an emphasis to clinical outcome parameters and further response assessments (e.g. peripheral immunmonitoring, imaging parameters) To prospectively assess patient-reported outcome of MEB patients To evaluate compliance to MEB suggestions in routine clinical care

ELIGIBILITY:
Inclusion Criteria:

* Chronic inflammatory disorder (PsO, PsA, SpA, IBD)
* Given informed consent
* 18 years of age

Exclusion Criteria:

* No capacity to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic inflammatory diseases and indication for therapy with biologic agents
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Therapy persistence | Through study completion, an average of 1 year
  Duration of intervention with biological agent

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tübingen - Center for Personalized Medicine, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided